CLINICAL TRIAL: NCT05665205
Title: Benefits of an Aerobic and Strength Rehabilitation Program With Post-SARS-CoV-2 Patients Moderate-severe
Brief Title: Benefits of an Aerobic and Strength Rehabilitation Program With Post- SARS-CoV-2 Patients Moderate-severe
Acronym: SARS-CoV-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, David Fernández, Benefits of an aerobic and strength program with Post-SARS-CoV-2 patients moderate-severe, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COV_2022
Record Dates: First submitted 2022-12-22; First posted 2022-12-27 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: Rehabilitation; COVID; Strenght exercise; Aerobic program
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Main investigators will be masked based on a randomization program. Outcomes Assessors will be not aware of the enrollment of participants and the study design to guaranty blinding of themselves.
  Participants will be randomized by a program and they will not be aware about which groups could be more beneficial to guarantee blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise plus strength (Active Comparator): The purpose is to verify if the aerobic exercise plus a strength program improves more than aerobic exercise alone in COVID patients.
  Interventions: Other: Aerobic plus strength group
- Aerobic exercise alone (Sham Comparator): The purpose is to verify if COVID patients can improve the status of their health only with an aerobic exercise program alone.
  Interventions: Other: Aerobic group

INTERVENTIONS:
Other: Aerobic plus strength group — A 8 week program of aerobic exercise plus strength exercise of upper and lower limbs in the hospital with a supervised trained physiotherapist
  Arms: Aerobic exercise plus strength
Other: Aerobic group — This group has a 8 weeks program of only aerobic exercise in the hospital with a supervised trained physiotherapist.
  Arms: Aerobic exercise alone

SUMMARY:
The SARS-CoV-2 is a pulmonary pathology which is caused by SARS-COV2 and the main signs and symptoms are fever, dyspnea, cough, fatigue, muscular pain and more. Even if SARS-CoV-2 is an acute respiratory pathology we know that can cause some chronic conditions in the general status health of the patients. Besides, it can have an important impact in the physique condition such as a detrimental of the aerobic capacity, lung capacity based on the severity of the patient.

On the other hand, World Health Organization (WHO) has a criteria to classify the severity of SARS-CoV-2;

Saturation de O2 <94%,

PaO2/FiO2: <300mm

Frecuencia respiratoria > 30p/m

abscess Lung > 50%

septic shock

Multiorganic failure

Based on the high survival but the important number of side effects of this pathology remaining the detrimental of the health and exercise condition. We justify our study based on an aerobic exercise program with a strength part to improve those conditions of the patients.

DETAILED DESCRIPTION:
The investigators develop an aerobic exercise program for two treatment groups which one of them has a strength program as a supplement to verify if the aerobic exercise plus strength improve more than aerobic exercise alone the condition of COVID patients.

The protocol is based on 8 weeks of program with a baseline measurements and a follow ups after the 8º weeks, at 2, 4 and six months after finish the treatment to compare the effectiveness of both treatment and between them.

ELIGIBILITY:
Inclusion Criteria:

* Patients had been got covid in the last 2 years.
* No fractures, or major injuries which could compromised the movements of the patient
* No major pathologies which deteriorate the general health status

Exclusion Criteria:

* Psychiatric (moderate to severe)
* Acute infection
* Fractures (moderate to severe)
* Cognitive detrimental state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
6MWT | 6 minutes
  The 6-minute walking test (6MWT) measured the cardiovascular endurance and the Functional Independence Measure assessed the global functional capacity
sf 36 | 36 minutes
  The 36-Item Short Form Health Survey (SF-36) is a widely it. The measure meets high psychometric standards [20, 21]. The 36 items represent eight scales: Physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health. These eight scales form two higher order constructs: physical health (the first four scales) and mental health (the latter four scales). These constructs are represented by two summary measures: Physical Component Summary (PCS) measure and Mental Component Summary (MCS) measure. Scoring was completed as per standard instructions, using norm-based scoring algorithms. Lower scores on the MCS refect "frequent psychological distress, substantial social and role disability due to emotional problems; health in general rated 'poor'". Lower scores on the PCS refect "Substantial limitations in self-care, physical, social, and role activities; severe bodily pain; frequent tiredness; health rated 'poor'"
Timed up and Go (TUG) | 5-7 minutes
  Functional mobility was assessed through the timed up-and-go (TUG) test, five times sit-to-stand (FTSTS) test, functional reach and balance confidence. The TUG test measures the time taken by a participant to stand from a sitting position, walk 3 m, return and sit back down and is a measure of mobility. The FTSTS measures the time taken by a participant to switch from sitting-to-standing five times in a row and is a test of functional strength. Functional reach measures the distance a participant can reach forward with his or her arm outstretched while standing and is a test of balance. For each test, participants completed a practice run before the actual measurement

SECONDARY OUTCOMES:
BORG | 10 seconds
  it is a scale that has been used to evaluate the degree of dyspnea (0=no dyspnea, 10=worse dyspnea)
Ecography | 2-3 minutes
  quadriceps muscle length will be measured
Heart beat | 45 min
  the heart beat will be measured before and during the treatment sessions
Saturation | 45 min
  Before the session and during the itself will be measured
SARC-F questionnaire | 10 minutes
  SARC-F includes five components: strength, assistance walking, rise from a chair, climb stairs, and falls. SARC-F items were selected to reflect health status changes associated with the consequences of sarcopenia. SARC-F scale scores range from 0 to 10 (i.e. 0-2 points for each component; 0 = best to 10 = worst) and were dichotomized to represent symptomatic (4+) vs. healthy (0-3) status

CONTACTS AND LOCATIONS:
Overall Officials: David Fernández, msc, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Locations (1):
- David Fernández, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
When the study will be completed and published, It will be available to share with more researches.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available at the end of the last follow up to have all data for the Statistical analysis.
Access Criteria: All data Access will be possible when the manuscript will be published in a Journal.

REFERENCES:
- [Background] Bohannon RW, Crouch R. 1-Minute Sit-to-Stand Test: SYSTEMATIC REVIEW OF PROCEDURES, PERFORMANCE, AND CLINIMETRIC PROPERTIES. J Cardiopulm Rehabil Prev. 2019 Jan;39(1):2-8. doi: 10.1097/HCR.0000000000000336. PMID 30489442
- [Background] Vilagut G, Valderas JM, Ferrer M, Garin O, Lopez-Garcia E, Alonso J. [Interpretation of SF-36 and SF-12 questionnaires in Spain: physical and mental components]. Med Clin (Barc). 2008 May 24;130(19):726-35. doi: 10.1157/13121076. Spanish. PMID 18570798